CLINICAL TRIAL: NCT04794283
Title: Antenatal Hand Milking for Pregnant Women With Diabetes
Brief Title: Antenatal Hand Milking for Pregnant Women With Diabetes'
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Other Study IDs: 2020-06042
Record Dates: First submitted 2021-03-01; First posted 2021-03-12 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Type 1; Diabetes Mellitus, Type 2; GDM
Keywords: Diabetes type1; Diabetes type2; GDM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Milk, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hand milking with Diabetes: 93 women with DM1, DM2 and medically treated GDM who are patients in specialist maternity care at Soderhospital in Stockholm and who plan to hand milk are part of this group.
  Interventions: Other: Breast milk
- Not hand milking with diabetes: A group of 93 women are then selected from 1 April 2021and back in the same number as the group1 (n=93) this group only gave milk substitute the first 24h.

INTERVENTIONS:
Other: Breast milk — Milk substitute given during the first 24h
  Other Names: Milksubstitute
  Groups: Hand milking with Diabetes

SUMMARY:
The project is a descriptive cohort study with a retrospective and a prospective group where pregnancy and childbirth data will be studied. Mothers with DM1, DM2, GDM hand-milk 2 times/day from v.36+0, freeze the colostrum they receive and bring it to delivery ward. The colostrum will then be given instead of milk substitutes for their children postpartum.

The primary questions are whether there is any statistical difference between a group that provides only colostrum compared to an equal retrospective group, which has only been given milk substitutes, in the case of neonatal hypoglycemia in the first 24 hours postpartum.

Secondly: 10 healthy women and 10women with DM1 will provide analysis of colostrum at week 36 of pregnancy. The secondary question is if there is any differences in colostrum whether the mother is healthy or has DMtype1

DETAILED DESCRIPTION:
The project is a descriptive cohort study with a retrospective and a prospective group where pregnancy and childbirth data will be studied. 93 mothers with DM1, DM2, GDM will hand-milk 2 times/day from v.36+0, freeze the colostrum they receive and bring it to delivery ward. The colostrum will then be given instead of milk substitutes for their children postpartum.

Population: 93 women with DM1, DM2 and medically treated GDM who are patients in specialist maternity care at Soderhospital in Stockholm, and who plan to hand milk, are the prospective group. A retrospective group of 93 diabetic women is then selected from 1 April 2021 and back from the medical database used in the clinic and they represent the retrospective group where milk substitutes has been given.

The primary question of the study is whether there is any statistical difference between a group of diabetic newborn that provides only colostrum compared to an equal retrospective group, which has only given milk substitutes, in the case of neonatal hypoglycemia in the first 24 hours postpartum.

Second question in the study is to study the difference in developing sun-treatment-demanding icterus between the children who received colostrum or milk substitutes first 24h and possible transfer of them to neonatal care.

Maternal outcome and background data will be retrieved from the maternal medical files.

The woman's diabetes status will also be retrieved: what type of diabetes, duration of diabetes, blood sugar levels + Hba1c values and possibly treatment (insulin and/or metformin).

Delivery data such as: Labor onset ( spontaneous, induction, cesarean sectio). Progress and outcome (normal delivery, VE, sectio). Oxytocin stimulation. Pain relief.

Information about the newborn like: - Gestational age at birth. Gender, Height and weight. Apgar scores at 1', 5' and 10' min. - The child's blood sugar levels during the first 24 hours (at least three occasions). Number of occasions of hypoglycemia in the child in the first 24 hours (limit value <2.6 mmol/L).

* Bilirubin values and possible sun treatment of the child.
* Possible transfer of the child to the neonatal ward, and its cause,
* If the child has been fed with milk substitute and if so with what.

As the second part of the project, breast milk from 10 of the pregnant women with DM1, included in the prospective group, as well as 10 pregnant women who do not have diabetes will be asked for participation in that part of the study aimed to analyzing the content of colostrum.

The study participants will hand-milk at least 10ml of colostrum at pregnancy weeks 36, 37, 38, 39, 40, 41, 42 and freeze it and she will take all the milk in a freezer-clad cooler when she goes into childbirth. At postpartum days 1, 2, 3, 4 and 5, breast milk will also be collected. After that, the raw milk contains are analyzed on:

* Fats
* Proteins
* Calories
* Carbohydrates
* Total Solids Any differences between the two groups will be presented in logistical regressions.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women with DM1, DM2 and medically treated GDM

Women must:

1. Be patients in specialist maternity care at the hospital
2. Plan to hand milk during pregnancy
3. Start at 36w of gestation

Exclusion Criteria:

* women who don't have diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women with diabetes
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
neonatal hypoglycemia on day 0 of life will be meassured | day 0
  The child's blood sugar levels in the first day of life (at least three occasions).
  - the number of occasions of hypoglycemia in the child in the first 24 hours (limit value <2,6 mmol/L),

SECONDARY OUTCOMES:
Hyperbilirubinemia during the first week of life will be meassured | First week of life
  High Bilirubin values within the first week of life

CONTACTS AND LOCATIONS:
Overall Officials: Eva Wiberg-Itzel, Profeesor, Principal Investigator — Karolinska Institutet
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monemi E, Tingstrom J, Sterpu I, Wiberg-Itzel E. The impact of lowering the blood glucose cut-off values in gestational diabetes mellitus on maternal and perinatal outcomes. Eur J Obstet Gynecol Reprod Biol. 2025 Apr;307:43-48. doi: 10.1016/j.ejogrb.2025.01.031. Epub 2025 Jan 22. PMID 39889557